CLINICAL TRIAL: NCT00526812
Title: A Phase I Dose-finding and Pharmacokinetic Study of Intravenous RTA 744 Injection in Patients With Recurrent or Refractory Anaplastic Astrocytoma (AA), Anaplastic Oligodendroglioma (AO), Anaplastic Mixed Oligo-astrocytoma (AOA), Glioblastoma Multiforme (GBM) or Gliosarcoma (GS), With or Without Concurrent Treatment With Enzyme-inducing Anticonvulsant Therapy
Brief Title: A Safety Study of RTA 744 in Patients With Recurrent High-Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTA 744-C-0401; NCT00346203 (obsolete NCT alias)
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — WP 744

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (RTA 744) (Experimental): Receive study drug for three consecutive days, Cycle repeated every 21 days.
  Interventions: Drug: RTA 744
- Group C (RTA 744 Injection) (Experimental): Receive study drug once a week for four consecutive weeks. Repeat cycle every 5 weeks.
  Interventions: Drug: RTA 744 injection

INTERVENTIONS:
Drug: RTA 744 — Aqueous solution added to 10%D/W and infused over 2 hours on three consecutive days. 5 mg vials contain 1 mg/ml.
  Arms: Group A (RTA 744)
Drug: RTA 744 injection — Aqueous solution in 1mg/ml. Doses are escalated. Drug is infused intravenously over 2 hours one day a week for four consecutive weeks.
  Arms: Group C (RTA 744 Injection)

SUMMARY:
This study assesses the tolerability, safety, efficacy and pharmacokinetics of RTA 744 in recurrent high-grade gliomas.

DETAILED DESCRIPTION:
Malignant gliomas, glioblastoma multiforme and anaplastic astrocytoma, are rapidly growing primary brain tumors associated with a high degree of morbidity and mortality. Despite aggressive treatment, the median survival rate for GBM is approximately 12 months, with two-year survival rates no more than 8 to 12%, while median survival for patients with AA ranges from 2 to 3 years from time of first diagnosis.

RTA 744 is a close chemical analogue of the well characterized anti-cancer agent doxorubicin. Unlike doxorubicin, RTA 744 has shown ability to cross the blood brain barrier and to achieve high concentration in CNS tumor tissue in animal models. It will be administered by i.v. infusions either daily for 3 consecutive days repeated every three weeks, or once weekly for 4 consecutive weeks repeated every 5 weeks. Once the maximum tolerated dose is determined , a new group of patients will be enrolled into the study to evaluate the tolerability and MTD when administered on an expanded schedule (once a week).

ELIGIBILITY:
Inclusion Criteria:

* Prior histologically confirmed anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed oligo-astrocytoma, glioblastoma multiforme, or gliosarcoma, for whom no other effective therapy is available.
* A prior histologic diagnosis of a lower grade of glioma is allowed if there is current histologic proof of progression to a diagnosis of AA, AO, AOA, GBM or GS
* Unequivocal evidence of recurrence or progression by neuroimaging procedure.
* Surgical resection at least 2 weeks prior to enrollment and must have completely recovered from the side effects.
* A stable dose of steroids for at least 7 days prior to obtaining the Gd-MRI of the brain.
* Previously implanted Gliadel® wafer may be eligible.
* Karnofsky Performance Status (KPS) of ≥ 60.
* Laboratory parameters: Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L, Hemoglobin (Hgb) ≥ 9 g/dl, Platelets ≥ 100 x 109/L, AST and ALT ≤ 3.0 x Upper Limit of Normal (ULN), Serum bilirubin ≤ 1.5 x ULN, Serum creatinine ≤ 1.5 x ULN and 24 hour creatinine clearance ≥ 50 ml/min
* Life expectancy of greater than 12 weeks.
* Written informed consent obtained.

Exclusion Criteria:

* Pregnancy or breast feeding, or adults of reproductive potential not employing an effective method of birth control
* Total urinary protein in 24 hours urine collection > 500 mg
* Any concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study.
* Impaired cardiac function, other significant prior cardiac disease or arrhythmia of any
* A history of CHF or arrhythmias.
* Therapeutic doses of warfarin sodium (Coumadin®).
* Prior or concurrent therapy, or not recovered from the toxic effects of such therapy: investigational drugs, chemotherapy, metronomic daily dosing of chemotherapy agents, biologic, immunotherapy or cytostatic agents within 4 weeks prior to study entry; radiation therapy within 2 weeks prior to study entry, any medication known to cause QT interval prolongation
* Any surgery other than resection of a brain tumor within 2 weeks prior to enrollment.
* A contraindication to MRI imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-11-30 (Actual); Primary Completion 2008-12-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of RTA 744 Injection in the patient population studied and to determine the qualitative and quantitative toxic effects of RTA 744 Injection. | at end of first cycle for each patient cohort

SECONDARY OUTCOMES:
To characterize the multiple-dose pharmacokinetics of RTA 744 and to document any potential antitumor activity of RTA 744 in those patients with measurable disease. | end of study

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA School of Medicine, Department of Neurology, Los Angeles, California
  - Baylor University Medical Center: Neuro-Oncology Associates, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/